CLINICAL TRIAL: NCT06020924
Title: The Effects of Uterine Fibroids on Pregnancy in Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wenwen Wang (Other)
Collaborators: Huazhong University of Science and Technology (Other); Shandong University (Other); Peking University People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Wenwen Wang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: UF1.0
Record Dates: First submitted 2023-06-22; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Female Infertility; Uterine Fibroid
Keywords: Infertility; Uterine fibroids; Pregnancy rate
MeSH Terms: conditions — Infertility, Female; Leiomyoma; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UFs with infertile patients: Uterine fibroids combined with infertile women
  Interventions: Other: No intervention
- UFs with non-infertile patients: Uterine fibroids combined with non-infertile women
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This study is a retrospective observational study without intervention.

SUMMARY:
Female fertility may be affected by uterine fibroids, although this association has not been elucidated. This retrospective cohort study aims to evaluate the impact of fibroids on women fertility.

DETAILED DESCRIPTION:
Infertility is defined as the inability of a couple to achieve pregnancy over an average period of one year of unprotected sexual intercourse. Currently, one in six couples is affected by infertility worldwide. With the development of society bringing enormous material and spiritual wealth to human beings, comprehensive factors such as environmental pollution, life and work pressure and bad habits have an important impact on fertility. Infertility is a disease that seriously affects the physical and mental health of patients and brings about serious social problems. According to the World Health Organization (WHO), infertility will become the third major disease in the 21st century following tumor and cardiovascular diseases.

Infertility can be caused by a single factor or multiple factors together. The WHO proposed a classification method based on etiological diagnosis to classify infertility into six major causes: ovulation factors, fallopian tube problems, uterine factors, cervical factors, male factors and psychosocial factors. There is a serious impact on female fertility due to heredity, auto-immunity, infection, metabolic abnormalities, surgery and other factors. The main factors leading to female infertility include patient age, education level, weight (obesity), menstrual history (irregular menstrual cycle), pregnancy history (stillbirth and abortion history), disease history (ovarian cyst, ovarian aging, endocrine autoimmune diseases, fallopian tube abnormalities, pelvic abnormalities and uterine abnormalities), sexual history, previous surgical history, smoking history, chemical exposure history, and mental stress, etc. The objective of this study is to explore the impact of uterine fibroids on female pregnancy rate.

Uterine fibroid is a common benign tumor of female reproductive tract, with 25% to 50% of women of childbearing age suffering from uterine fibroid. The fibroids can cause various clinical symptoms, including menorrhagia, prolonged menstruation, pelvic compression and pain, as well as infertility and obstetric complications, but mostly are asymptomatic. The prevalence of fibroids increases with the age of women, while the fertility rate declines with ages. This complex relationship is particularly harmful. The mechanisms related to fibroids and infertility vary with the type and location of fibroids, including anatomical structure deformation, and interference with the physiological changes of endometrium and implantation of zygotes. In addition, fibroids can destroy the anatomical structure of the pelvis and disrupt the function of the fallopian tube. The FIGO classification describes nine types of fibroids: submucosal fibroids (type 0, Ⅰ, Ⅱ), intramural fibroids (types Ⅲ, Ⅳ, Ⅴ), and subserous fibroids (types Ⅵ and Ⅶ). Among them, submucosal and some intramural fibroids can lead to endometrial inflammatory environment, affecting sperm migration and embryo implantation.

Nevertheless, there is still controversy in epidemiological studies regarding the relationship between uterine fibroids and female infertility. Parity has a significant protective effect against fibroid development, and in fact infertile women may be at higher risk for fibroids. Similarly, it is difficult to distinguish whether fibroids have a direct deleterious effect on infertility, or whether the fibroid-infertility association is mediated by concomitant factors that affect fertility. In addition, the impact of each type of fibroids on fertility varies by the difference in the number, size, and location of fibroids, and the combinations of different fibroids may have special effects. Do uterine fibroids already exist when women plan and attempt to conceive? Do uterine fibroids have negative effects on fertility during this period? It is an urgent need to solve this problem at the present. Therefore, this study is of great significance for us to understand the impact of fibroids on female fertility and guide the treatment patterns of female patients with uterine fibroids who have fertility needs.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-50 years
2. Diagnosed with uterine fibroids (by ultrasound or pathology) combined with infertile or non-infertile patients
3. Complete clinical data.

Exclusion Criteria:

1. Severe infectious disease or rheumatic immune disease active stage
2. Previous history of malignant tumors
3. Incomplete clinical data.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female patients with uterine fibroids
Sampling Method: Non-Probability Sample
Enrollment: 1658 (Estimated)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The pregnancy rate varies with different types and size of fibroids. | through study completion, an average of 2.5 year
  Fibroid types range from 0 to 8 according to the FIGO classification. The pregnancy rate varies with different types and size of fibroids. Subserosal fibroids do not exert any detrimental effects on fertility outcomes. Submucosal fibroids have negatively impact fertility. The effect of intramural fibroids on reproductive outcome has been a subject of debate in the past, but recent literature indicates that intramural myomas also negative impact fertility.

SECONDARY OUTCOMES:
The rate of spontaneous abortion varies with different types and size of fibroids. | through study completion, an average of 2.5 year
  Fibroids are a source of several obstetric complications, including spontaneous abortion, preterm birth, cesarean section, placental abruption, postpartum hemorrhage, and breech presentation. Submucosal fibroids and multiple myomas have an increased risk of miscarriage. The rate is calculated as the proportion of the number of miscarriage to the total number of pregnancies in different types of fibroids.
The rate of preterm birth varies with different types and size of fibroids. | through study completion, an average of 2.5 year
  Fibroids measuring more than 5 centimetre (cm) have been linked to delivery at earlier gestational age. The ratio is calculated as the proportion of fibroids combined with preterm birth to fibroids combined with live birth.
The rate of cesarean section varies with different types and size of fibroids. | through study completion, an average of 2.5 year
  Greater size and number of fibroids were associated with increased incidence of cesarean delivery. The ratio is calculated as the proportion of fibroids combined with cesarean section to total births.
The rate of placental abruption varies with different types and size of fibroids. | through study completion, an average of 2.5 year
  Fibroids have an increased risk of placental abruption in patients. The ratio is calculated as the proportion of fibroids combined with placental abruption to total patients.
The rate of postpartum hemorrhage varies with different types and size of fibroids. | through study completion, an average of 2.5 year
  There is an independent association of uterine leiomyomata with increased risk of severe postpartum hemorrhage. Submucosal fibroids are less implicated in bleeding events than intramural and subserosal ones. Great rates of hemorrhage are related with the biggest lesions. The ratio is calculated as the proportion of fibroids combined with postpartum hemorrhage to total patients.
The rate of malpresentation varies with different types and size of fibroids. | through study completion, an average of 2.5 year
  Patients with fibroids have an increased risk of breech presentation. Malpresentation may be more related to multiple fibroids an to those bigger than 10 cm. The ratio is calculated as the proportion of fibroids combined with malpresentation to total patients.

CONTACTS AND LOCATIONS:
Overall Officials: Shixuan Wang, Principal Investigator — Huazhong University of Science and Technology, Wuhan, Hubei, China, 430000
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No